CLINICAL TRIAL: NCT02829697
Title: The Effect of Local Anaesthetic Volume on Nerve Block Duration and Nerve Block Duration Variability. A Randomised, Blinded, Healthy Volunteer Study
Brief Title: The Effect of Local Anaesthetic Volume on Nerve Block Duration and Nerve Block Duration Variability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Claus Behrend Christiansen, MD, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-16000184
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Pain
Keywords: Regional anaesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Peroneal nerve: Ropivacaine 0.2%, 2.5 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 2,5 mL
  Interventions: Drug: Ropivacaine
- Peroneal nerve: Ropivacaine 0.2%, 5 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 5 mL
  Interventions: Drug: Ropivacaine
- Peroneal nerve: Ropivacaine 0.2%, 10 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 10 mL
  Interventions: Drug: Ropivacaine
- Peroneal nerve: Ropivacaine 0.2%, 15 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 15 mL
  Interventions: Drug: Ropivacaine
- Peroneal nerve: Ropivacaine 0.2%, 20 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 20 mL
  Interventions: Drug: Ropivacaine
- Sciatic nerve: Ropivacaine 0.2%, 5 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 5 mL
  Interventions: Drug: Ropivacaine
- Sciatic nerve: Ropivacaine 0.2%, 10 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 10 mL
  Interventions: Drug: Ropivacaine
- Sciatic nerve: Ropivacaine 0.2%, 15 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 15 mL
  Interventions: Drug: Ropivacaine
- Sciatic nerve: Ropivacaine 0.2%, 20 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 20 mL
  Interventions: Drug: Ropivacaine
- Sciatic nerve: Ropivacaine 0.2%, 30 mL (Active Comparator): Perineural injection of ropivacaine 0.2 %, 30 mL
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Perineural injection.

SUMMARY:
The aim is to investigate the effect of perineural administration of a series of different volumes of local anaesthesia (ropivacaine 0.2%) on nerve block duration and the variability of the duration in the common peroneal nerve and the sciatic nerve in healthy volunteers.

The hypothesis is that nerve block duration is correlated to local anaesthetic volume, but only to a certain degree. After a sufficient volume a 'saturation level' will be reached, and nerve block duration will not increase further.

DETAILED DESCRIPTION:
The trial is divided into two similar phases. Each phase will focus on a specific nerve. Phase 1 will focus on the common peroneal nerve and Phase 2 will focus on the sciatic nerve.

After baseline measurements, the investigators will insert a peripheral intravenous catheter. Then, the investigators will insert a suture-method peripheral nerve catheter (Certa CatheterTM). Procedures will be done in a sterile manner as a standard of practice. The investigators will use an ultrasound (US)-guided short-axis, needle in-plane technique. For the US-scan, the investigators will use a linear or a curvilinear transducer.

During interventions, volunteers will be monitored with continuous pulse oximetry. Placement of the peripheral nerve catheter will be facilitated by US using small injections of mepivacaine (carbocaine 2 %) in the skin and surrounding tissues and only isotonic saline (5 mL) in the perineural space to prevent blocking of the nerve before ropivacaine injection. The catheter orifice will be placed by pulling either end of the catheter and guided by the built-in echogenic markings seen on US. Before injection of ropivacaine, the investigators will do careful aspirations through the catheter in order to prevent intravasal injection.

Each ropivacaine injection will be administered via an infusion pump. This will ensure a constant infusion rate set to 10 mL per minute. During infusion, the volunteers will be monitored with continuous pulse oximetry.

Before instigation of the ropivacaine infusion, the investigators will use US to verify full absorption of the isotonic saline in the perineural space.

For each nerve, the subject will be randomly allocated to and receive one of five possible ropivacaine volumes. All volunteers and outcome assessors will be blinded to the ropivacaine administrations and infusion procedures. Outcome assessors will not be in the room, when the medication is prepared nor given. Preparation will take place behind a curtain and therefore also blinded to the volunteers.

ELIGIBILITY:
Inclusion criteria

1. Male or female 18-64 years
2. American Society of Anesthesiologists Classification ≤ II

Exclusion criteria

1. Body Mass Index ≤ 18 or ≥ 30
2. Former surgery to the lower extremities
3. Peripheral nerve disease
4. Allergy to ropivacaine
5. Pregnancy or breastfeeding
6. Enrolment in other investigational drug studies or recent clinical trials that may interfere with this study
7. Habitual use of any kind of analgesic treatment
8. Anatomic abnormalities preventing successful US-guided peripheral nerve catheter insertion

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Duration of sensory nerve block | 1-24 hours
  Application of a round, cooled glass container in the sensory distribution area of the tested nerve: The lateral part of the lower leg for the common peroneal nerve and beneath the foot for the tibial nerve. Testing will start after onset of sensory nerve block and continue until normal sensation has returned. When testing the sciatic nerve, we will continue testing until normal sensation has returned in both components of the nerve, i.e. the tibial and common peroneal nerve.

SECONDARY OUTCOMES:
Length of nerve exposed to local anaesthesia | 10 minutes
  We will measure local anaesthetic spread in a proximal-to-distal manner parallel to the nerve trajectory. Total length of the neural spread will be reported in millimetres from the most proximal point to the most distal point in which fluid, i.e. ropivacaine, is seen on ultrasound in proximity to the nerve. Testing will be done immediately after end of ropivacaine infusion.
Onset of sensory nerve block | 10-180 minutes
  Application of a round, cooled glass container in the sensory distribution area of the tested nerve: The lateral part of the lower leg for the common peroneal nerve and beneath the foot for the tibial nerve. Testing will start ten minutes after end of infusion and continue for every fifth minute until onset. We will test for a maximum of 180 minutes.
Onset of motor nerve block | 10-180 minutes
  Testing will start ten minutes after end of infusion and continue for every fifth minute until onset. When onset of sensory nerve block is confirmed, testing of motor nerve block onset will end as well, if not already found. Motor nerve block of the tibial nerve will be evaluated by plantarflexion of the ankle. Motor nerve block of the common peroneal nerve will be tested by dorsiflexion of the ankle.
Degree of sensory nerve block | 1-24 hours
  We will test sensory nerve block using a subjective rating scale. We will grade from one to four: 1) "not different from ipsilateral antebrachium"; 2) "different from ipsilateral antebrachium"; 3) "warm sensation"; 4) "no sensation". Grades 2-4 will be considered as successful sensory nerve blocks. It will be noted if the volunteer is in doubt. Nevertheless, this will be considered as a successful sensory nerve block and graded as 2) in the post hoc statistical analyses.
Degree of motor nerve block | 1-24 hours
  This will be tested with the volunteer in the upright position using a sturdy counter for balance if necessary. Motor strength will be evaluated using a normal everyday activation of the lower leg: A toe and a heel raise, testing the common peroneal nerve via activation of the anterior tibial muscle and the tibial nerve via activation of the gastrocnemius muscle, respectively. Motor nerve block intensity will be evaluated on a scale from one to three: 1) normal strength, 2) paresis or 3) paralysis. Volunteers will be asked to perform a maximum contraction building up muscle force over three seconds. It will be noted if the volunteer is in doubt, which will be considered as 2) paresis in the post hoc statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Henrik Wiborg Lange, MD DMSC, Study Director — Nordsjællands Hospital Hillerød
Locations (1):
- Claus Behrend Christiansen, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We will attach relevant data sheets to all our scientific submissions.